CLINICAL TRIAL: NCT03925064
Title: Fetal Myocardial Performance Index in Diabetic Pregnancies
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.7.06
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-04

CONDITIONS: Gestational Diabetes; Myocardial Dysfunction
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic pregnancies: Pregnant women with pregestational or gestational diabetes mellitus
  Interventions: Other: myocardial performance index
- non-diabetic pregnancies: Pregnant women without pregestational or gestational diabetes mellitus
  Interventions: Other: myocardial performance index

INTERVENTIONS:
Other: myocardial performance index — fetal right ventricular myocardial performance index measured with tissue doppler

SUMMARY:
The myocardial tissue is the most likely structure affected by hyperglycemia. The myocardial performance index (MPI) is a pulsed wave Doppler-derived index of global myocardial function. It is defined as the sum of the isovolumetric contraction time (ICT) and isovolumetric relaxation time (IRT) divided by the ejection time (ET) The fetal right heart contributes more to the cardiac output than the left heart; therefore, it is important to assess the right ventricular function. The investigators will measure right ventricular MPI in diabetic and normal pregnancies.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is the most common metabolic disorder in pregnancy, with an overall prevalence of 3-7 % during pregnancy. The myocardial tissue is the most likely structure affected by hyperglycemia. The myocardial performance index (MPI) is a pulsed wave Doppler-derived index of global myocardial function. It is defined as the sum of the isovolumetric contraction time (ICT) and isovolumetric relaxation time (IRT) divided by the ejection time (ET) The fetal right heart contributes more to the cardiac output than the left heart; therefore, it is important to assess the right ventricular function. The investigators will measure right ventricular MPI in diabetic and normal pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old pregnant women

Exclusion Criteria:

* fetal cardiac anomalies
* multiple gestations

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 18-40 years old pregestational or gestational diabetic women
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
ultrasonographic myocardial performance index values | during procedure
  cardiac contractility will be measured with Doppler ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSRTH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No